CLINICAL TRIAL: NCT02207829
Title: A Randomized, Blinded, Double-dummy, Parallel-group Study to Evaluate the Efficacy and Safety of Umeclidinium (UMEC) 62.5 mcg Compared With Tiotropium 18 mcg in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 12-week Study to Evaluate the Efficacy and Safety of Umeclidinium Compared With Tiotropium in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201316
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; inhaler critical errors; double-dummy; novel dry powder inhaler; inhaler preference; tiotropium; umeclidinium; long-acting muscarinic antagonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium 62.5 mcg + placebo (Experimental): Subjects will receive UMEC Inhalation Powder 62.5 mcg once daily via nDPI plus placebo once daily via HANDIHALER inhaler for 12 weeks (24 weeks in Germany). Subjects will be instructed to take one inhalation each morning from both the nDPI and the HANDIHALER inhaler
  Interventions: Drug: Umeclidinium; Drug: Umeclidinium matching placebo
- Tiotropium 18mcg + placebo (Active Comparator): Subjects will receive Tiotropium 18 mcg once daily via HANDIHALER inhaler plus placebo once daily via nDPI for 12 weeks (24 weeks in Germany). Subjects will be instructed to take one inhalation each morning from both the nDPI and the HANDIHALER inhaler
  Interventions: Drug: Tiotropium; Drug: Tiotropium matching placebo

INTERVENTIONS:
Drug: Umeclidinium — Umeclidinium 62.5 mcg once daily in the morning via nDPI
  Arms: Umeclidinium 62.5 mcg + placebo
Drug: Umeclidinium matching placebo — Umeclidinium matching placebo once daily in the morning via nDPI
  Arms: Umeclidinium 62.5 mcg + placebo
Drug: Tiotropium — Tiotropium 18 mcg once daily in the morning via HANDIHALER inhaler
  Arms: Tiotropium 18mcg + placebo
Drug: Tiotropium matching placebo — Tiotropium matching placebo once daily in the morning via HANDIHALER inhaler
  Arms: Tiotropium 18mcg + placebo

SUMMARY:
This is a multicentre, randomized, blinded, double dummy, parallel group study to evaluate the efficacy and safety of UMEC inhalation powder[ (62.5 microgram (mcg) once daily (QD)] when administered via a novel Dry Powder Inhaler compared with tiotropium (18 mcg QD) administered via a HANDIHALER® inhaler over a treatment period of 12 weeks (24 weeks in Germany) in subjects with chronic obstructive pulmonary disease (COPD). At the end of the run-in period, subjects who meet the randomization criteria will be randomized to receive UMEC 62.5 mcg administered via novel dry powder inhaler(nDPI) + Placebo administered via HANDIHALER inhaler OR Tiotropium 18 mcg administered via HANDIHALER inhaler + Placebo administered via nDPI in a 1:1 ratio. There will be up to 8 clinic visits conducted on an outpatient basis at Pre-Screening (Visit 0), Screening (Visit 1), a 7 to 14 day run-in period, randomization at Day 1 (Visit 2), and after randomization at Day 2 (Visit 3), Day 28 (Visit 4), Day 56 (Visit 5), Day 84 (Visit 6) and Day 85 (Visit 7). For subjects enrolled in Germany, there will be an additional 3 visits at Day 112 (Visit 8), Day 140 (Visit 9) and Day 168 (Visit 10). The total duration of subject participation in the study will be approximately 15 weeks (27 weeks in Germany). The primary endpoint of the study is clinic visit trough forced expiratory volume in one second (FEV1) on treatment Day 85. All subjects will have spirometry performed at clinic Visits 1 though 7. Trough spirometry will be obtained 23 and 24 hours after the previous day's dose of blinded study medication at Visits 3 to 7.

HANDIHALER is a registered trademark of Boehringer Ingelheim Pharma GmbH & Co. KG.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male and female subjects are eligible to participate in the study. A female is eligible to enter and participate in the study if she is of:

Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, > 45 years, in the absence of hormone replacement therapy. OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact). - Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society

* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g. 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack-years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack-year history.
* Severity of Disease: A pre and post-albuterol/salbutamol FEV1/ Forced Vital Capacity (FVC) ratio of <0.70 and a post-albuterol/salbutamol FEV1 of >=30% and <=70% of predicted normal values at Visit 1. Predicted values will be based upon the ERS Global Lung Function Initiative
* Dyspnea: A score of >=2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known Alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other Diseases/Abnormalities: Any subject who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g. cancer). In addition, any subject who has any condition (e.g. neurological condition) that is likely to affect respiratory function should not be included in the study.
* Severe Hepatic Impairment: Patients with severe hepatic impairment (Child-Pugh class C) should be excluded unless, in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Moderate to severe Renal Impairment: Patients with moderate to severe renal impairment (e.g., end-stage renal disease requiring dialysis) should be excluded, unless in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Unstable or life threatening cardiac disease: Long-acting muscarinic antagonists (LAMAs) should be used with caution in subjects with severe cardiovascular disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association Class IV heart failure
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, sympathomimetic, lactose/milk protein or magnesium stearate.
* Antimuscarinic effects: Subjects with medical conditions such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction should only be included if, in the opinion of the study physician, the benefit outweighs the risk.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead electrocardiogram (ECG): Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. Subjects with the following abnormalities are excluded from participation in the study: Atrial fibrillation with rapid ventricular rate >120 beats per minute; Sustained or nonsustained ventricular tachycardia; Second degree heart block Mobitz type II or third degree heart block (unless pacemaker or defibrillator had been inserted)
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids-12 weeks; Systemic, oral or parenteral corticosteroids- 6 weeks; Antibiotics (for lower respiratory tract infection)- 6 weeks ; long-acting beta2-agonists/inhaled corticosteroids (LABA/ICS) combination products if LABA/ICS therapy is discontinued completely-30 days; LABA/ICS combination products only If discontinuing ICS/LABA therapy and switching to ICS monotherapy- 48 hours for the salmeterol or formoterol component, 14 days for the vilanterol component [The dose of ICS must be a dose of fluticasone propionate (FP) or equivalent but not to exceed 1000 mcg/day] ; Use of ICS at a dose >1000 mcg/day of FP or equivalent- 30 days; Initiation or discontinuation of ICS use-30 days (Use of ICS is permitted provided the dose does not exceed 1000mcg of FP or equivalent; ICS use not to be initiated or discontinued within 30 days prior to Visit 1, except for subjects on LABA/ICS therapy who may discontinue the ICS/LABA product as indicated in the table above and switch to ICS monotherapy); Phosphodiesterase 4 (PDE4) Inhibitor (roflumilast)- 14 days; Inhaled long acting beta2 agonists (LABAs): salmeterol, formoterol-48 hours, olodaterol, indacaterol, vilanterol- 14 days; LAMAs: tiotropium, aclidinium, glycopyrronium, umeclidinium- 7 days; LAMA/LABA combination products if LAMA/LABA therapy is discontinued completely- Apply whichever mono component has the longest washout; Theophyllines- 48 hours; Oral beta2-agonists: Long-acting- 48 hours, Short-acting 12 hours; Inhaled short acting beta2-agonists- 4 hours (Use of study provided albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing) ; Inhaled short-acting anticholinergics- 4 hours; Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products- 4 hours; Any other investigational medication - 30 days or within 5 drug half lives (whichever is longer).
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e. <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g. albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or write would not be able to complete a questionnaire

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1017 (Actual)
Dates: Start 2014-09-01; Primary Completion 2015-05-25 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (81):
- GSK Investigational Site, Spartanburg, South Carolina, United States
- GSK Investigational Site, Buenos Aires, Argentina
- Canada (9):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Chile (3):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talcahuano
- Denmark (4):
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Odense
- France (5):
  - GSK Investigational Site, Bletterans
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vieux-Condé
- Germany (9):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Rodgau, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
- Italy (5):
  - GSK Investigational Site, Riccione (RN), Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Torrette (AN), The Marches
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Negrar, Veneto
- Romania (10):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Comuna Alexandru Cel Bun
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Focşani
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Russia (14):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Sestroretsk
  - GSK Investigational Site, Sochi
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Vladimir
- South Africa (10):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Boksburg, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Korsten
  - GSK Investigational Site, Lynnwood Ridge, Pretoria
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Vrededorp
  - GSK Investigational Site, Welkom
- South Korea (3):
  - GSK Investigational Site, Bucheon-Si, Gyeonggi-Do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wonju-si, Gangwon-do
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kryvyi Rig
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Shah D, Driessen M, Risebrough N, Baker T, Naya I, Briggs A, Ismaila AS. Cost-effectiveness of umeclidinium compared with tiotropium and glycopyrronium as monotherapy for chronic obstructive pulmonary disease: a UK perspective. Cost Eff Resour Alloc. 2018 May 10;16:17. doi: 10.1186/s12962-018-0101-3. eCollection 2018. PMID 29773969
- [Derived] Feldman G, Maltais F, Khindri S, Vahdati-Bolouri M, Church A, Fahy WA, Trivedi R. A randomized, blinded study to evaluate the efficacy and safety of umeclidinium 62.5 mug compared with tiotropium 18 mug in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2016 Apr 7;11:719-30. doi: 10.2147/COPD.S102494. eCollection 2016. PMID 27103795
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (Par.), with clinical history of chronic obstructive pulmonary disease, who met eligibility criteria at screening were enrolled in a 7 to 14 days run-in period. Eligible par. were randomized (1:1) to receive umeclidinium or tiotropium. A total of 1214 par. were screened; 1017 par. were randomized and entered into the study.
Groups:
- Umeclidinium 62.5 mcg+Placebo QD: Participants received umeclidinium (UMEC) inhalation powder 62.5 microgram (mcg) once-daily (QD) in morning via a novel dry powder inhaler (nDPI) and placebo QD via alternative dry powder inhaler (DPI) for 12 weeks (For participants enrolled in Germany, the duration of treatment was 24 weeks). Participants also received albuterol/salbutamol via metered-dose-inhaler (MDI) or nebules as rescue medication throughout the study for use as needed.
- Tiotropium 18 mcg+Placebo QD: Participants received tiotropium (TIO) 18 mcg QD in morning via DPI and placebo QD via nDPI for 12 weeks (For participants enrolled in Germany, the duration of treatment was 24 weeks). Participants also received albuterol/salbutamol via MDI or nebules as rescue medication throughout the study for use as needed.
Period: Overall Study
Arm/Group | Umeclidinium 62.5 mcg+Placebo QD | Tiotropium 18 mcg+Placebo QD
Started | 509 | 508
Completed | 467 | 474
Not Completed | 42 | 34
Not completed — Adverse Event | 10 | 9
Not completed — Lack of Efficacy | 7 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol deviation | 5 | 4
Not completed — Withdrew consent | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umeclidinium 62.5 mcg+Placebo QD | Tiotropium 18 mcg+Placebo QD | Total
Number analyzed (Participants) | 509 | 508 | 1017
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.12) | 64.1 (8.28) | 64.2 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 137 | 282
  Male | 364 | 371 | 735
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 9 | 9 | 18
  American Indian or Alaska Native | 1 | 0 | 1
  Central/South Asian Heritage | 0 | 1 | 1
  Japanese/East Asian/South East Asian Heritage | 38 | 37 | 75
  White | 458 | 457 | 915
  African American/African Heritage & White | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) on Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Day 84 (Week 12). Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84 and 85. Baseline trough FEV1 is the mean of the two assessments made -30 and -5 minutes (min) pre-dose on Day 1. Change from baseline was calculated as the trough FEV1 value on Day 85 minus the BL value. Analysis performed using a repeated measures model with covariates of treatment, baseline FEV1, centre group, 24 hour subset flag, Day, Day by baseline and Day by treatment interactions. The least squares mean changes are presented here.
Time Frame: Baseline (BL) and Day 85
Population: Per Protocol(PP) Population(pop): Participants(par) in the Intent-To-Treat pop who did not have a full protocol deviation considered to impact efficacy. Par represent those with data available at time point presented; however, all par. in the PP pop. without missing covariate information and >=1 post BL measurement are included in analysis
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Umeclidinium 62.5 mcg+Placebo QD | Tiotropium 18 mcg+Placebo QD
Number analyzed (Participants) | 392 | 416
Liter | 0.154 (0.0107) | 0.095 (0.0106)
Statistical Analysis 1: Comparison: Umeclidinium 62.5 mcg+Placebo QD vs Tiotropium 18 mcg+Placebo QD; Test type: Non-Inferiority or Equivalence — Alternate hypothesis: the difference between the trt means (umeclidinium minus tiotropium) would be > -50 milliliters (mL). If the lower CI (2.5% 1-sided significance level) of the statistical test should fall above -50 mL, then umeclidinium may be deemed statistically non-inferior to tiotropium. If the lower CI (2.5% 1-sided significance) of the statistical testing exceeded 0 then, umeclidinium may be deemed statistically superior to tiotropium; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [0.029 to 0.088]

ADVERSE EVENTS:
Time Frame: On-treatment(trt) non-serious adverse events(AEs) and serious AEs are events occurring while par were on trt or events with an onset during follow-up period(up to 13 weeks). AE data for German subjects are only included for the first 12 weeks of trt.
Description: On-treatment non-serious AEs and SAEs were reported for the ITT Population comprised all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | Umeclidinium 62.5 mcg+Placebo QD | Tiotropium 18 mcg+Placebo QD
Serious Adverse Events (participants affected / at risk) | 17/509 | 16/508
Other Adverse Events (participants affected / at risk) | 50/509 | 52/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Umeclidinium 62.5 mcg+Placebo QD (N=509) | Tiotropium 18 mcg+Placebo QD (N=508)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airway disease (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Umeclidinium 62.5 mcg+Placebo QD (N=509) | Tiotropium 18 mcg+Placebo QD (N=508)
Headache (Nervous system disorders) | 30 | 32
Nasopharyngitis (Infections and infestations) | 27 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.